CLINICAL TRIAL: NCT07141329
Title: An Open-Label Extension, One-Year, Safety, and Efficacy Study of SPN-817 in Adults With Focal Onset Seizures
Brief Title: SPN-817 Open-Label Extension Study in Adults With Focal Onset Seizures
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Supernus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 817P210
Record Dates: First submitted 2025-08-19; First posted 2025-08-26 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Focal Onset Seizures
Keywords: focal seizures; focal epilepsy; open-label extension; anti-seizure medication
MeSH Terms: conditions — Seizures; Epilepsies, Partial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SPN-817 (Experimental): SPN-817, bid
  Interventions: Drug: SPN-817

INTERVENTIONS:
Drug: SPN-817 — SPN-817 starting at 0.25 mg bid up to 4.00 mg bid

SUMMARY:
This is a Phase 2b open-label extension study to evaluate the long-term safety and efficacy of SPN-817.

DETAILED DESCRIPTION:
This is a Phase 2b, multicenter, open-label extension, one-year, safety, tolerability, and efficacy study in adults who previously completed an applicable double-blind SPN-817 clinical study. This study will include a double-blind Dose Titration/Bridging Period of 8-10 weeks in which SPN-817 will be titrated to the participant's maximum tolerated dose based on response. Following the Dose Titration/Bridging Period, participants will enter an Open Label Extension (OLE) Period of 42-44 weeks. When participants finish the OLE Period, they will initiate a Tapering Period (up to 4 weeks) followed by an End-of-Tapering Period video contact (VC) after the last dose of study drug. The duration of study treatment before starting the 4-week Tapering Period will be one year (52 weeks).

ELIGIBILITY:
Inclusion Criteria:

1. Completed antecedent SPN-817 double-blind study
2. Taking a stable dosage regimen (maintained during the antecedent study) of at least one antiseizure medication (ASM) and no more than 4 ASMs

Exclusion Criteria:

1. Has current nonepileptic events that could be confused by the participant and/or study staff as epileptic seizures
2. Has any suicidal behavior or suicidal ideation related to Item 4 (active suicidal ideation with some intent to act without specific plan) or Item 5 (active suicidal ideation with specific plan and intent) based on the Columbia-Suicide Severity Rating Scale (C-SSRS) assessments in the antecedent study and at Visit 1 or more than one lifetime suicide attempt.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | Week 1-Week 52
  The percent of participants who took at least one dose of SPN-817 and reported at least one adverse event during the 1-year SPN-817 Treatment Period

SECONDARY OUTCOMES:
Percent change (PCH) from baseline in quantifiable focal onset seizure frequency per 28 days over the 1-year SPN-817 Treatment Period | Baseline and Treatment Period (Week 1-52)
  Percent change in 28-day frequency of quantifiable focal seizures during the 1-year Treatment Period relative to baseline
Proportion of participants experiencing ≥50% reduction in focal seizure frequency per 28 days from baseline | Baseline and Treatment Period (Week 1-52)
  Greater than or equal to 50% reduction in 28-day frequency of focal seizures during the 1-year Treatment Period relative to baseline.
Proportion of participants experiencing seizure freedom | Baseline and Treatment Period (Week 1-52)
  100% reduction in 28-day frequency of focal seizures during the Treatment Period relative to baseline
Percentage of seizure-free days over the 1-year SPN-817 Treatment Period | Week 1-Week 52
  The number of seizure-free days reported for each participant divided by the total number of days with seizure data reported, multiplied by 100.

CONTACTS AND LOCATIONS:
Overall Officials: Maciej Gasior, MD, PhD, Study Director — Supernus Pharmaceuticals, Inc.
Locations (1):
- Medsol Clinical Research Center, Port Charlotte, Florida, United States